CLINICAL TRIAL: NCT03260595
Title: A Phase 1, Single-center, Randomized, Vehicle-controlled, Parallel-cohort Study Of Crisaborole Ointment 2% To Evaluate The Skin Irritation Potential In Adult Japanese Healthy Subjects, And To Evaluate The Safety, Tolerability And Pharmacokinetics In Adult Japanese Subjects With Mild To Moderate Atopic Dermatitis
Brief Title: A Study of Crisaborole Ointment 2% in Adult Japanese Healthy Subjects and Adult Japanese Subjects With Mild To Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: C3291029
Record Dates: First submitted 2017-08-09; First posted 2017-08-24 (Actual); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Healthy; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisaborole ointment 2% (Experimental)
  Interventions: Drug: Crisaborole ointment 2%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Crisaborole ointment 2% — Crisaborole ointment 2%
  Arms: Crisaborole ointment 2%
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
This is a Phase 1 parallel-cohort study of crisaborole ointment 2% to evaluate the skin irritation potential in adult Japanese healthy subjects in Cohort 1, and to evaluate the safety, tolerability and PK in adult Japanese subjects with mild to moderate AD in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

1. Healthy male Japanese subjects who, at the time of screening, are between the ages of 20 and 55 years, inclusive.
2. Healthy skin on which reddening can be easily recognized in the area of the test fields.

Cohort 2

1. Male or female Japanese subjects aged 20 years to 55 years (inclusive) at the time of screening, and in generally good health except for AD.
2. Diagnosis of AD based on the criteria of Hanifin and Rajka (1980).
3. Has at least 25% Treatable %BSA on Day 1 (excluding the scalp and designated venous access areas).
4. Has an Investigator's static global assessment (ISGA) score of Mild (2) or Moderate (3) on Day 1.

Exclusion Criteria:

Cohort 1

1. Subjects who have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction.
2. Subjects who have psoriasis and/or active AD/eczema.
3. Subjects who have a history of AD.
4. Subjects who have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site.
5. Known sensitivity to any of the components of the investigational products.
6. History of the rash to the adhesive plaster, contact dermatitis to metal, or cosmetic and household articles.

Cohort 2

1. Has any clinically significant medical disorder, condition, disease (including active or potentially recurrent dermatological conditions other than AD), significant physical examination or laboratory findings that may interfere with study objectives, in the Investigator's opinion.
2. Has unstable AD or a consistent requirement for strong to strongest potency topical corticosteroids to manage AD signs and symptoms.
3. Has a significant active systemic or localized infection, including known actively infected AD.
4. Has a history or evidence of clinically significant or severe allergies (eg, seasonal, pet dander, environmental, food) requiring acute or chronic treatment.
5. Has recent or anticipated concomitant use of topical or systemic therapies that might alter the course of AD.
6. Has a history of recent (within 4 weeks of Day 1) sunbathing, tanning bed use, or ultraviolet (UV) light B therapy (UVB) or psoralen plus UVA [PUVA]).
7. Has a known sensitivity to any of the components of crisaborole ointment 2%.
8. Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3291029&StudyName=A+Phase+1%2C+Single-center%2C+Randomized%2C+Vehicle-controlled%2C+Parallel-cohort+Study+Of+Crisaborole+Ointment+2%25+To+Evaluate+The+Skin+Irritation+Potential+In+Adult+Japanese+Healthy+Subjects%2C+And+To+Evaluate+The+Safety%2C+Tolerability+And+Pharmacokinetics+In+Adult+Japanese+Subjects+With+Mild+To+Moderate+Atopic+Dermatitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Crisaborole Ointment 2% and Vehicle: Crisaborole ointment 2 percent (%) and matching vehicle was applied topically to 2 randomly assigned, adjacent sites on the skin area field at infrascapular area of the back respectively within each healthy participant under occlusive patch condition on Day 1. Ointment and vehicle were remained under occlusion for 48 hours. Target sites were identified at Baseline (Day 1) by investigator.
- Cohort 2: Crisaborole Ointment 2%: Crisaborole ointment 2% was applied topically to the treatable percent body surface area (%BSA: defined as percent of a participant's total BSA that is atopic dermatitis [AD]-involved and is not on the scalp or in designated venous access areas) of participants with AD twice daily from Days 2 to 7 and once only on Days 1 and 8. Treatable %BSA was calculated at Baseline (Day 1) by investigator.
- Cohort 2: Vehicle: Vehicle matched to Crisaborole ointment 2% was applied topically to the treatable %BSA (defined as percent of a participant's total BSA that AD-involved and is not on the scalp or in designated venous access areas) of participants with AD twice daily from Days 2 to 7 and once only on Days 1 and 8. Treatable %BSA was calculated at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | Cohort 1: Crisaborole Ointment 2% and Vehicle | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
Started | 20 | 10 | 2
Completed | 20 | 10 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least one dose of study medication.
Groups:
- Cohort 1: Crisaborole Ointment 2% and Vehicle: Crisaborole ointment 2% and matching vehicle was applied topically to 2 randomly assigned, adjacent sites on the skin area field at infrascapular area of the back respectively within each healthy participant under occlusive patch condition on Day 1. Ointment and vehicle were remained under occlusion for 48 hours. Target sites were identified at Baseline (Day 1) by investigator.
- Cohort 2: Crisaborole Ointment 2%: Crisaborole ointment 2% was applied topically to the treatable percent body surface area (%BSA: defined as percent of a participant's total BSA that is AD-involved and is not on the scalp or in designated venous access areas) of participants with AD twice daily from Days 2 to 7 and once only on Days 1 and 8. Treatable %BSA was calculated at Baseline (Day 1) by investigator.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Crisaborole Ointment 2% and Vehicle | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle | Total
Number analyzed (Participants) | 20 | 10 | 2 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.66) | 35.0 (11.28) | 23.5 (4.95) | 28.8 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 10 | 2 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 2 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 10 | 2 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Skin Irritation Index
Description: The skin irritation index is a common measure of skin irritation potential (safety criteria) of investigational product and derived using skin irritation scores. Individual skin irritation score ranges from 0-4, where 0 = no reaction, 0.5 = mild erythema, 1 = erythema, 2 = erythema with edema and papula, 3 = erythema with edema, papula and small water blister, 4 = large water blister, higher score indicates more skin irritation. For each investigational product, the skin irritation index was calculated as the sum of the maximum individual skin irritation scores divided by the number of evaluable participants and multiplied by 100, which ranged from 0 to 400; where, lower score indicated less skin irritation and higher score indicated more skin irritation.
Time Frame: Day 3 to 4
Population: Safety analysis population included all participants who received at least one dose of study medication. Data for this outcome measure was not planned to be collected and analyzed for Cohort 2, as pre-specified in protocol.
Measure: Number; unit: scores on a scale
Arm/Group | Cohort 1: Crisaborole Ointment 2% and Vehicle
Number analyzed (Participants) | 20
scores on a scale
  Crisaborole ointment 2% | 40.0
  Vehicle | 5.0

2. Primary Outcome: Cohort 2: Number of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose of study drug (up to Day 36) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to Day 36
Population: Safety analysis population included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
Number analyzed (Participants) | 10 | 2
Participants
  AEs | 9 | 2
  SAEs | 0 | 0

3. Primary Outcome: Cohort 2: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included pulse rate and blood pressure. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to end of treatment (Day 8)
Population: Safety analysis population included all participants who received at least one dose of study medication. Data for this outcome measure was not planned to be collected and analyzed for Cohort 1, as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
Number analyzed (Participants) | 10 | 2
Participants | 0 | 0

4. Primary Outcome: Cohort 2: Number of Participants With Laboratory Tests Abnormalities
Description: Laboratory tests abnormalities included: hematology (haemoglobin[Hb], haematocrit and erythrocytes<0.8*lower limit of normal[LLN]; erythrocyte mean corpuscular volume, erythrocyte mean corpuscular Hb and erythrocyte mean corpuscular Hb concentration <0.9*LLN and >1.1*upper limit of normal[ULN]; platelets <0.5*LLN and >1.75*ULN; leukocytes <0.6*LLN and >1.5*ULN; lymphocytes/leukocytes[%], neutrophils/leukocytes[%] <0.8*LLN and >1.2*ULN; basophils/leukocytes[%], eosinophils/leukocytes[%], monocytes/leukocytes[% ]>1.2*ULN); clinical chemistry(bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase>3.0*ULN; protein and albumin<0.8*LLN and >1.2*ULN; urea nitrogen and creatinine >1.3*ULN; urate>1.2*ULN; sodium <0.95*LLN and >1.05*ULN; potassium, chloride and calcium <0.9*LLN and >1.1*ULN; fasting glucose <0.6*LLN and >1.5*ULN); and urinalysis (pH <4.5 and >8; glucose, ketones, protein, Hb, urobilinogen, bilirubin, nitrite and leukocyte esterase >=1).
Time Frame: Baseline up to end of treatment (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
Number analyzed (Participants) | 10 | 2
Participants | 7 | 1

5. Primary Outcome: Cohort 2: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant ECG abnormalities included: QT interval >=500 milliseconds (msec); QT interval corrected using the Fridericia's formula (QTcF) >=450 msec to <480 msec, >=480 msec and >=500 msec; increase from baseline in QTcF interval >=30 msec to <60 msec and >=60 msec.
Time Frame: Baseline up to end of treatment (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
Number analyzed (Participants) | 10 | 2
Participants | 0 | 0

6. Secondary Outcome: Cohort 1: Number of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose of study drug (up to Day 29) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to Day 29
Population: Safety analysis population included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Crisaborole Ointment 2% and Vehicle
Number analyzed (Participants) | 20
Participants
  AEs | 0
  SAEs | 0

7. Secondary Outcome: Cohort 2: Maximum Observed Plasma Concentration (Cmax) of Crisaborole and Its Identified Main Oxidative Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and Day 8
Population: PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. Data for this outcome measure was not planned to be collected and analyzed for Cohort 1, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
nanograms per milliliter (ng/mL)
  Crisaborole: Day 1 | 163.7 (71)
  Crisaborole: Day 8 | 164.9 (56)
  AN7602: Day 1 | 94.97 (75)
  AN7602: Day 8 | 68.83 (59)
  AN8323: Day 1 | 3064 (97)
  AN8323: Day 8 | 8080 (71)

8. Secondary Outcome: Cohort 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crisaborole and Its Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and Day 8
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
hours
  Crisaborole: Day 1 | 3.000 [3.00 to 3.00]
  Crisaborole: Day 8 | 3.000 [3.00 to 3.00]
  AN7602: Day 1 | 3.000 [3.00 to 3.00]
  AN7602: Day 8 | 3.000 [3.00 to 3.00]
  AN8323: Day 1 | 3.000 [3.00 to 12.0]
  AN8323: Day 8 | 3.000 [3.00 to 12.0]

9. Secondary Outcome: Cohort 2: Area Under the Plasma Concentration-Time Curve From Time Zero Until the Last Measurable Concentration (AUClast) of Crisaborole and Its Identified Main Oxidative Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter(hr*ng/mL)
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
hours*nanograms per milliliter(hr*ng/mL)
  Crisaborole: Day 1 | 1171 (60)
  Crisaborole: Day 8 | 1527 (48)
  AN7602: Day 1 | 601.9 (60)
  AN7602: Day 8 | 565.5 (44)
  AN8323: Day 1 | 57560 (84)
  AN8323: Day 8 | 169100 (68)

10. Secondary Outcome: Cohort 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the 24 Hours Post-Dose (AUC24) of Crisaborole and Its Identified Main Oxidative Metabolites (AN7602 and AN8323)
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
hr*ng/mL
  Crisaborole: Day 1 | 1171 (60)
  Crisaborole: Day 8 | 1527 (48)
  AN7602: Day 1 | 601.9 (60)
  AN7602: Day 8 | 565.5 (44)
  AN8323: Day 1 | 57560 (84)
  AN8323: Day 8 | 169100 (68)

11. Secondary Outcome: Cohort 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Tau (12 Hours Dosing Interval) (AUCtau) of Crisaborole and Its Identified Main Oxidative Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole. AUC tau was defined as area under the plasma concentration-time curve from time 0 to time tau, the dosing interval, where tau =12 hours.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
hr*ng/mL
  Crisaborole: Day 1 | 928.9 (65)
  Crisaborole: Day 8 | 1123 (51)
  AN7602: Day 1 | 500.4 (66)
  AN7602: Day 8 | 434.9 (50)
  AN8323: Day 1 | 29360 (92)
  AN8323: Day 8 | 90360 (68)

12. Secondary Outcome: Cohort 2: Accumulation Ratio for Cmax (Rac [Cmax]) of Crisaborole and Its Identified Main Oxidative Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole. Accumulation ratio for Cmax (Rac, Cmax) was calculated as Cmax on Day 8 divided by Cmax on Day 1. Cmax was the maximum plasma concentration of Crisaborole and its identified main oxidative metabolites.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
ratio
  Crisaborole | 1.007 (32)
  AN7602 | 0.7247 (24)
  AN8323 | 2.638 (52)

13. Secondary Outcome: Cohort 2: Accumulation Ratio for AUCtau (Rac [AUCtau]) of Crisaborole and Its Identified Main Oxidative Metabolites
Description: AN7602 and AN8323 were the main identified oxidative metabolites of Crisaborole. Accumulation ratio for AUCtau (Rac) was calculated as area under the curve from time zero to end of dosing interval (AUCtau) on Day 8 divided by AUCtau on Day 1. Dosing interval = 12 hours.
Time Frame: Pre-dose, 3, 12 and 24 hours post-dose on Day 1 and 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2: Crisaborole Ointment 2%
Number analyzed (Participants) | 9
ratio
  Crisaborole | 1.209 (25)
  AN7602 | 0.8688 (19)
  AN8323 | 3.080 (48)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29 for Cohort 1 and Day 36 for Cohort 2
Arm/Group | Cohort 1: Crisaborole Ointment 2% and Vehicle | Cohort 2: Crisaborole Ointment 2% | Cohort 2: Vehicle
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 0/20 | 9/10 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Crisaborole Ointment 2% and Vehicle (N=20) | Cohort 2: Crisaborole Ointment 2% (N=10) | Cohort 2: Vehicle (N=2)
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Application site coldness (General disorders) | 0 | 1 | 1
Application site irritation (General disorders) | 0 | 7 | 1
Application site pain (General disorders) | 0 | 4 | 1
Application site pruritus (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03260595/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03260595/SAP_001.pdf